CLINICAL TRIAL: NCT03139357
Title: Behavioral Monitoring in Primary Care
Status: Terminated | Type: Observational
Why Stopped: Tech changes made it impossible to consent patients. Not a flaw in design, practice changes caused the study end.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eva Szigethy, Professor of Psychiatry, University of Pittsburgh
Other Study IDs: 16090557
Record Dates: First submitted 2017-01-25; First posted 2017-05-03 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Life Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary care patients: Patients ages 20-65 who score 5 or greater on the GAD-7 will be given the SF12, GAD7, medial utilization, and helpfulness questionnaires at 6 month intervals for a 2 year period.
  Interventions: Other: GAD7, SF12, medical utilization, helpfulness questionnaire

INTERVENTIONS:
Other: GAD7, SF12, medical utilization, helpfulness questionnaire — The questionnaires are administered to track stress level and medical utilization over a 2 year period.

SUMMARY:
Stress and anxiety can worsen quality of life in patients seen in primary care practices. Patients at predetermined practices age 20-65 receive psychosocial screening instruments for anxiety and quality of life (GAD7 and SF-12) at six month intervals for twenty-four months as part of routine care. Assessing anxiety and quality of life every six months will provide data to analyze whether anxiety and quality of life changes over time.

Patients who consent will also be asked at 6, 12, 18, and 24 months about medical utilization of behavioral care or any medical care outside of University of Pittsburgh Medical Center in order to be part of their research record for good clinical care. If patients received any behavioral treatment, the patient will also be asked questions regarding the helpfulness of this treatment.

This is an observational characterization study to understand the psychiatric and behavioral needs of primary care patients. The follow-up questionnaires and medical record information will look at the rates and predictors of hospitalizations and/ or behavioral health treatment as a longitudinal way to track these symptoms over time. These resources are critical to determine the need for embedded behavioral care in primary care settings.

DETAILED DESCRIPTION:
Patients who are receiving or seeking medical care at University of Pittsburgh Medical Center CMI practices are given the GAD7(anxiety) and SF-12(quality of life) as a part of routine medical care. Patient scores become part of the EMR (Epic). A best practice alert will be generated for patients in the age range of 20-65 (inclusive) and in the targeted GAD7 score range (GAD7 ≥5) to prompt the provider to obtain consent. Within 2-4 weeks after consent, a UPMC research team member will administer via phone a brief, approximately 10 minute questionnaire for patients who score ≥10 on the GAD7 questionnaire and have signed consent. This DSM5 cross-cutting measure level 1 is a validated screening tool capturing primary psychiatric symptoms present across a range of disorders. A secure database will be maintained within the UPMC firewall where all patient information will be de-identified. Routine care safety protocols are in place if a patient's anxiety/stress worsens. At 6,12,18, and 24 months post-consent, the research team will contact the patient by phone to complete routine questionnaires (GAD7 and SF-12) if questionnaires have not been completed in clinic at an appointment or via the patient portal, MyUPMC. As part of the study, the patient will complete the Medical Utilization/Follow up questionnaire by phone with the research team at the 6, 12, 18, and 24 month time points. If the patient had any behavioral health treatment the research team will also ask the Helpfulness Questionnaire at the six month time point. In addition to these questionnaires, the research team will access Epic records to understand medical utilization.

CARe will provide the information from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* receiving or seeking medical care at UPMC CMI
* ages 20-65
* GAD7 (anxiety questionnaire) score ≥ 5
* Speaks English speaking
* Capable of understanding and providing consent or assent

Exclusion Criteria:

* under age 20 and older than 65
* GAD7 score <5
* patients with acute back pain

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ages 20-65 at designated UPMC primary care sites who score 5 or greater on the GAD7 (anxiety) questionnaire. This questionnaire is given as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
GAD7 score change over time | 2 years (6, 12, 18, 24 months)
  mesures anxiety

SECONDARY OUTCOMES:
SF-12 score change over time | 2 years (6, 12, 18, 24 months)
  measures quality of life
Medical hospitalization days change over time | 2 years (6, 12, 18, 24 months)
  measures medical utilization as number of days inpatient
ER visits change over time | 2 years (6, 12, 18, 24 months)
  measures medical utilization as number of visits to the emergency dept.
Outpatient clinic visits change over time | 2 years (6, 12, 18, 24 months)
  measures medical utilization as number of PCP clinic visits
Number of phone calls to practice change over time | 2 years (6, 12, 18, 24 months)
  Phone call from subject to PCP practice

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, MD PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided